CLINICAL TRIAL: NCT05185843
Title: An Open-Label Safety Study of AKCEA-APOCIII-LRX Administered Subcutaneously to Patients With Familial Chylomicronemia Syndrome (FCS) Previously Treated With Volanesorsen (ISIS 304801)
Brief Title: A Study of Olezarsen (Formerly Known as AKCEA-APOCIII-LRX) Administered to Adults With Familial Chylomicronemia Syndrome (FCS) Previously Treated With Volanesorsen
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Ionis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ISIS 678354-CS7; 2021-003635-29 (EudraCT Number); 2023-508815-22-00 (EU CTIS Number)
Expanded Access: NCT06360237 (Approved for marketing)
Record Dates: First submitted 2021-11-20; First posted 2022-01-11 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Familial Chylomicronemia Syndrome
Keywords: FCS
MeSH Terms: conditions — Familial hyperchylomicronemia syndrome | interventions — olezarsen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Olezarsen (Experimental): Olezarsen will be administered once every 4 weeks by subcutaneous (SC) injection for up to 209 weeks.
  Interventions: Drug: Olezarsen

INTERVENTIONS:
Drug: Olezarsen — Olezarsen will be administered by SC injection.
  Other Names: ISIS 678354; AKCEA-APOCIII-LRx

SUMMARY:
The purpose of the study is to evaluate the safety, tolerability, pharmacokinetic (PK) and pharmacodynamic (PD) effects of olezarsen (formerly known as AKCEA -APOCIII-LRX) in participants with FCS previously treated with volanesorsen.

DETAILED DESCRIPTION:
This is a Phase 3, multi-center, open-label safety study in 24 participants with FCS, previously treated with volanesorsen. The study consists of an 8- week screening period, treatment period up to week 209 and a 13-week follow-up period. Participants enrolled will receive olezarsen every 4 weeks during the 209-week Treatment Period.

Treatment period was extended to allow participants to receive olezarsen for an additional 52 weeks for a total of a 209-week treatment period until the drug may be commercially available in the patient's country, or until the Sponsor discontinues the olezarsen development program, whichever occurs earlier.

ELIGIBILITY:
Key Inclusion Criteria

1. Participants with FCS (clinical or genetic diagnosis) currently on or previously treated with volanesorsen (ISIS 304801)

   o Study participants in countries where Waylivra® is commercially approved and available for participants should not be deprived of the treatment option with Waylivra®. Participation in this study for such participants will only be allowed when Waylivra® was discontinued due to AEs
2. The following concomitant medications will be allowed if dosing regimen is expected to remain constant through the end of the study (occasional or intermittent use of over-the-counter (OTC) medications will be allowed at Investigator's discretion):

   * Statins, omega-3 fatty acids (prescription and OTC), fibrates, or other lipid-lowering medications. Participants taking OTC omega-3 fatty acids should make every effort to remain on the same brand through the end of the study
   * Antidiabetic medications
   * Oral anticoagulants (e.g., dabigatran, rivaroxaban, or apixaban, and warfarin with regular clinical monitoring)
   * Tamoxifen, estrogens or progestins

Key Exclusion Criteria:

1. Treatment with another investigational drug (non-oligonucleotide), biological agent, or device within 4 weeks of Screening, or 5 half-lives of investigational agent, whichever is longer
2. Concomitant medication/procedure restrictions:

   1. Systemic corticosteroids or anabolic steroids within 6 weeks prior to Screening and during the study unless approved by the Sponsor Medical Monitor
   2. Plasma apheresis within 4 weeks prior to Screening or planned during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-02-25 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Proportion of Participants With Decrease in Platelet Count by >30% or >50%, or With Platelet Count Value <50,000/cubic millimeter (mm^3) | Baseline to Week 209
Proportion of Participants With Clinical Bleeding Events | Baseline to Week 209
Proportion of Participants With Decrease in Estimated Glomerular Filtration Rate (eGFR) by ≥30% or ≥50% | Baseline to Week 209
Proportion of Participants With Urine Protein/Creatinine Ratio (UPCR) ≥1000 milligram (mg)/gram (g) or with Urine/Albumin Creatinine Ratio (UACR) ≥500 mg/g | Baseline to Week 209
Proportion of Participants With Alanine Aminotransferase (ALT) or Aspartate Aminotransferase (AST) ≥5 x Upper Limit of Normal (ULN) | Baseline to Week 209
Proportion of Participants With ALT or AST ≥3 x ULN and Total Bilirubin > 2 x ULN | Baseline to Week 209
Proportion of Participants With Total Bilirubin ≥2 mg/deciliter (dL) | Baseline to Week 209

SECONDARY OUTCOMES:
Trough (Pre-Dose) Plasma Concentration of Olezarsen | Up to 209 weeks
Post-Treatment Plasma Concentration of Olezarsen | Up to 209 weeks
Change and Percent Change From Baseline in Fasting Triglycerides (TG) | Baseline to Week 209
Change and Percent Change From Baseline in Fasting Apolipoprotein C-III (APOC-III) | Baseline to Week 209
Change and Percent Change From Baseline in Fasting Very Low-Density Lipoprotein (VLDL)-C | Baseline to Week 209
Change and Percent Change From Baseline in Fasting Chylomicron-TG | Baseline to Week 209
Change and Percent Change From Baseline in Fasting Total Cholesterol (TC) | Baseline to Week 209
Change and Percent Change From Baseline in Fasting Non-High-Density Lipoprotein (non-HDL)-C | Baseline to Week 209
Change and Percent Change From Baseline in Fasting Low-Density Lipoprotein (LDL)-C | Baseline to Week 209
Change and Percent Change From Baseline in Fasting Apoprotein B (apoB) | Baseline to Week 209
Change and Percent Change From Baseline in Fasting Apoprotein B48 (apoB48) | Baseline to Week 209
Change and Percent Change From Baseline in Fasting High-Density Lipoprotein (HDL)-C | Baseline to Week 209
Change and Percent Change From Baseline in Fasting Apoprotein A-1 (ApoA-1) | Baseline to Week 209
Event Rate of Acute Pancreatitis | Up to 209 weeks

CONTACTS AND LOCATIONS:
Locations (11):
- United States (4):
  - Diabetes/Lipid Management & Research Center, Huntington Beach, California
  - Excel Medical Clinical Trials, LLC, Boca Raton, Florida
  - University of Michigan, Department of Internal Medicine, Division of Metabolism, Endocrinology and Diabetes (MEND), Ann Arbor, Michigan
  - University of Rochester School of Medicine, Rochester, New York
- Canada (6):
  - Centre for Heart Lung Innovation, Vancouver, British Columbia
  - ARC Biosystems, Clinical Assessment Unit (CAU), Vancouver, British Columbia
  - St. Boniface General Hospital, Winnipeg, Manitoba
  - Ecogene-21, Chicoutimi, Quebec
  - Clinique des Maladies Lipidiques de Quebec Inc., Québec, Quebec
  - Centre Hospitalier Universite de Sherbrooke (CHUS), Sherbrooke, Quebec
- Karolinska University Hospital Huddinge, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Ionis may share anonymized individual participant data, aggregated clinical data, and other types of data that support the results in this study. Data requests from qualified researchers will be considered once all three of the following criteria are met: (1) 12 months from marketing approval of the study drug in both the United States and European Union; (2) 18 months from conclusion of the study; and (3) 6 months from publication of study article. Access would be via a secure environment and is contingent upon approval of a research proposal and entry into an appropriate data use agreement. Requests to access data can be submitted via the website https://vivli.org/ourmember/ionis/.
URL: https://vivli.org/ourmember/ionis/